CLINICAL TRIAL: NCT03251820
Title: Management Strategies for Electrical Status Epilepticus During Sleep
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Randa Abdelbadie Abdelaleem (Other)
Responsible Party: Sponsor-Investigator, Randa Abdelbadie Abdelaleem, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: MSESES
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy
Keywords: electrical status epilepticus during slow wave sleep; seizure; cognition; continuous spikes and waves during sleep
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: corticosteroid — Each patient will be subjected to a one month course of steroids and then re-evaluated

SUMMARY:
Electrical status epilepticus during slow wave sleep is a condition in which the epileptic patient starts to develop neurocognitive deterioration, any type of seizures and continuous electrical activity in the EEG during non rapid eye movement sleep. It is an age related condition and will resolve spontaneously at around the age of puberty. However if left untreated or treatment is delayed, it may lead to permanent neurocognitive deterioration. Thus early diagnosis and treatment is essential in these children to preserve neurocognitive function.

DETAILED DESCRIPTION:
Electrical status epilepticus in sleep (ESES), also known as continuous spikes and waves during slow sleep (CSWS), is an age related, self - limiting disorder characterized by:

1. epilepsy with different seizure types,
2. neuropsychological regression, and
3. typical EEG pattern of continuous epileptiform activity during non-rapid eye movement sleep (NREM).

During wakefulness, the EEG shows focal/multifocal spikes that increase in frequency during the acute stage. During sleep, ESES appears and is characterized by (1) marked potentiation of epileptiform discharges during non-REM sleep, leading to (2) a (near)-continuous, bilateral, or occasionally lateralized slow spikes and waves, (3) and these spikes and waves occur "during a significant proportion" of the non-REM sleep with a threshold ranging from 25% to 85%

The exact incidence of CSWS is not known. In pediatric neurology clinics, a reported frequency of 0.2% of childhood epilepsies most probably underestimates the incidence of CSWS.

CSWS is a devastating syndrome, which requires prompt treatment, the efficacy of which is checked with regular intervals, e.g. three or six months. Although epilepsy resolves with time in most cases, many children are left with significant cognitive or language impairment. Longer duration of ESES appears to be the major predictor of poor outcome.

So, early recognition and effective therapy are necessary to improve long-term prognosis in this condition.

The goal of treatment is not only to control clinical seizures but also to improve neuropsychological functions and prevent potential cognitive deterioration. There was no agreement on best treatment, but potential candidates included high-dose benzodiazepines, valproate, levetiracetam, and corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* All epileptic patients above 2 years of age presenting with neuropsychological deterioration, seizures and ESES in NREM sleep. The degree of epileptic activity during sleep will be measured and expressed as a spike wave index (SWI), which is defined as the total duration of continuous epileptic activity relative to total slow sleep duration. SWI must be at least 25% or more.

Exclusion Criteria:

* Any epileptic patient not presenting with typical EEG findings and neurocognitive regression.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Those patients who fulfill the inclusion criteria attending the neurology unit at Assiut University Children Hospital will be administered the following treatment: 1. Nocturnal diazepam for three months 2. Corticosteroids tapered over one months 3. Antiepileptic drug other than sodium channel blockers which will be continued for at least two years. During the course of the treatment the patients will be followed up by sleep EEG and IQ before and at least one month after the start of treatment and regularly every three months for at least one year after discontinuation of benzodiazepines and steroids.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive ability | IQ measured before treatment and after completing treatment course and then every three months for one year
  Change in cognitive ability in response to steroids and benzodiazepines by IQ assessment using using Standford - Binnet scales version V.
Interictal epileptiform activity | EEG will be done every three months for upto one year after discontinuation of therapy
  epileptiform activity will be assessed by EEG recordings during sleep. The degree of epileptic activity during sleep will be measured and expressed as a spike wave index (SWI), which is defined as the total duration of continuous epileptic activity relative to total slow sleep duration.

SECONDARY OUTCOMES:
Change in seizure frequency | Measured before and one year after treatment
  Compare the frequency of seizures before the start of treatment and after the start of treatment.